CLINICAL TRIAL: NCT06350006
Title: A Phase Ib/III Study of SHR-A1904 Combinations in CLDN18.2-Positive Advanced Solid Tumor
Brief Title: SHR-A1904 Combinations in CLDN18.2-Positive Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1904-301
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: CLDN18.2-positive Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: This study is a multicenter Phase Ib/III clinical study. Phase Ib consists of two stages, IB-A for dose escalation and IB-B for efficacy expansion. The Phase III multi-center, randomized ,active-controlled, Open-label study was designed to evaluate the efficacy and safety of SHR-A1904 combined chemotherapy and immunotherapy versus chemotherapy combined immunotherapy in first-line treatment of CLDN18.2-positive solid tumors patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1904 combined with Adebrelimab (Experimental): SHR-A1904+ Adebrelimab
  Interventions: Drug: SHR-A1904; Adebrelimab
- SHR-A1904 combined with CAPOX and Adebrelimab (Experimental): SHR-A1904+ CAPOX+ Adebrelimab
  Interventions: Drug: SHR-A1904; CAPOX; Adebrelimab

INTERVENTIONS:
Drug: SHR-A1904; Adebrelimab — SHR-A1904 combined with Adebrelimab: SHR-A1904+ Adebrelimab
  Arms: SHR-A1904 combined with Adebrelimab
Drug: SHR-A1904; CAPOX; Adebrelimab — SHR-A1904 combined with Adebrelimab and CAPOX (Capecitabine, Oxaliplatin)
  Arms: SHR-A1904 combined with CAPOX and Adebrelimab

SUMMARY:
This study consists of two research phases:

Phase Ib (includes dose escalation stage and efficacy expansion stage): To explore the safety, tolerability and initial efficacy of SHR-A1904 in the treatment of CLDN18.2-positive advanced solid tumors, and to determine the recommended dose and recommended population for the Phase III combination study.

Phase III: A randomized, Open-Label, multicenter clinical study of SHR-A1904 combined with chemotherapy and immunotherapy Versus chemotherapy combined with immunotherapy for CLDN18.2-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (including boundary values);
2. Volunteer to participate in this clinical study and sign informed consent;
3. ECOG score 0-1;
4. Expected survival ≥3 months;
5. Pathologically confirmed locally advanced unresectable or metastatic solid tumors;
6. positive CLDN18.2 expression in tumor tissue;
7. There is at least one measurable lesion that meets the RECIST 1.1 criteria;
8. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Plan to receive any other antitumor therapy during this trial; Received other investigational drugs or treatments that are not on the market within 4 weeks prior to the first administration; Anti-tumor therapy, such as chemotherapy, radiotherapy, biotherapy, targeted therapy or immunotherapy, was received within 4 weeks before the first administration of the study drug. Palliative radiotherapy or local therapy within 2 weeks before the first administration of the study drug; Had major surgery other than diagnosis or biopsy within the 4 weeks prior to the first administration or randomization and required elective surgery during the trial.
2. HER2 expression in tumor tissue is positive.
3. The adverse reactions of previous anti-tumor therapy has not recovered to NCI-CTCAE v5.0 grade≤ 1.
4. Has ≥ grade 2 peripheral sensory neuropathy.
5. Has an allergic reaction to any of the components treated in this study, or are allergic to humanized monoclonal antibody products.
6. Has a history or current history of meningeal metastasis; or active brain metastases.
7. Presence of dysphagia or other factors affecting the use of oral medications.
8. Additional malignancy within the five years prior to the first administration or randomization.
9. Has an active autoimmune disease or a history of autoimmune disease.
10. Received systemic use of corticosteroids or other immunosuppressants for immunosuppressive effects within 14 days prior to the first administration or randomization.
11. Has a history of clinically significant lung disease.
12. Has serosal effusion ≥ grade 3 (based on NCI CTCAE5.0 criteria).
13. There was an active infection requiring systemic treatment within 2 weeks prior to the first administration or randomization.
14. A history of immunodeficiency, including a positive HIV test; Presence of active hepatitis B or hepatitis C.
15. People who have previously received allogeneic hematopoietic stem cell transplantation or organ transplantation.
16. Has severe cardiovascular and cerebrovascular diseases.
17. Gastrointestinal perforation and/or gastrointestinal fistula within the last 6 months prior to the first administration or randomization; Active gastrointestinal bleeding occurred 3 months before the first administration or randomization.
18. In the investigator's judgment, the subject has other factors that could have affected the study results or led to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AE | Up to follow-up period, approximately 24 months
  Phase 1b
Dose Limiting Toxicity (DLT) | approximately 24 months
  Phase 1b
Maximal Tolerable Dose (MTD) | approximately 24 months
  Phase 1b
Phase III Recommended Dose (RP3D) | approximately 24 months
  Phase 1b
Progression-free survival (PFS) assessed by blind Independent Center Review (BICR) based on RECIST 1.1 criteria | approximately 36 months
  Phase 3

SECONDARY OUTCOMES:
SHR-A1904 toxin binding antibody | approximately 24 months
  Phase 1b
SHR-A1904 Total antibody | approximately 24 months
  Phase 1b
Immunogenicity indicators of SHR-A1904: drug resistant antibody (ADA) and neutralizing antibody (NAb) | approximately 24 months
  Phase 1b
Expression level of CLDN18.2 in tumor tissues | approximately 24 months
  Phase 1b
Overall survival (OS) | approximately 36 months
  Phase 3
Incidence and severity of AE | approximately 36 months
  Phase 3

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided